CLINICAL TRIAL: NCT01780987
Title: Active-control, Multicenter, Randomized, Open-label, Safety And Efficacy Study Evaluating The Use Of Apixaban In The Treatment Of Symptomatic Deep Vein Thrombosis And Pulmonary Embolism In Japanese
Brief Title: AStudy To Evaluate Safety And Eficacy Of Apixaban In Japanese Acute Deep Vein Thrombosis (DVT) And Pulmonary Embolism (PE) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0661024; CV185160 (Other: BMS)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: DVT; PE; VTE
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — apixaban; Heparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental)
  Interventions: Drug: Apixaban
- UFH/Warfarin (Active Comparator)
  Interventions: Drug: Unfractionated Heparin (UFH); Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban — 10 mg BID for 7 days followed by 5 mg BID for 23 weeks (total 24 weeks)
  Arms: Apixaban
Drug: Unfractionated Heparin (UFH) — Dosing adjustment based on APTT = 1.5-2.5 times the control value, and until INR ≥ 1.5 for 5 days or more
  Arms: UFH/Warfarin
Drug: Warfarin — Dosing for 24 weeks to target INR range between 1.5-2.5
  Arms: UFH/Warfarin

SUMMARY:
The purpose of this study is to investigate safety of apixaban in Japanese acute DVT/PE subjects when symptomatic DVT/PE subjects are treated with 10 mg BID apixaban for 7 days as initial therapy followed by 5 mg BID apixaban for 23 weeks as long-term therapy (total treatment period is 24 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Acute symptomatic proximal DVT with evidence of proximal thrombosis
* Acute symptomatic PE with evidence of thrombosis in segmental or more proximal branches

Exclusion Criteria:

* Active bleeding or high risk for bleeding contraindicating treatment with UFH and a VKA.
* Uncontrolled hypertension: systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg
* Subjects requiring dual anti-platelet therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Japan (20):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima General Hospital, Hatsukaichi, Hiroshima
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Kinki University Hospital, Sayama, Osaka
  - National Cerebral and Cardiovascular Center Hospital, Suita-shi, Osaka
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661024&StudyName=AStudy%20To%20Evaluate%20Safety%20And%20Eficacy%20Of%20Apixaban%20In%20Japanese%20Acute%20Deep%20Vein%20Thrombosis%20%28DVT%29%20And%20Pulmonary%20Embolism%20%28PE%29%20Patie

RESULTS

PARTICIPANT FLOW:
Groups:
- Apixaban: Two apixaban 5 mg tablets were administrated twice a day (morning and evening) for 7 days followed by one apixaban 5 mg tablet administrated twice a day (morning and evening) for 23 weeks.
- Unfractionated Heparin (UFH)/Warfarin: UFH was administrated by continuous intravenous infusion to bring the activated partial thromboplastin time (APTT) to between 1.5 and 2.5 times the control level, until the effect of warfarin stabilized. UFH was administrated at least 5 days unless international normalized ratio (INR) ≥ 2.0 was reached before Day 5. The appropriate dose of warfarin potassium to achieve the target INR range between 1.5 and 2.5 was administrated for 24 weeks.
Period: Overall Study
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Started | 40 | 40 (Including one participant who withdrew from the study prior to receiving any study medication.)
Completed | 37 | 34
Not Completed | 3 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Request of Changing Hospital | 0 | 1
Not completed — Changing Residence | 1 | 0
Not completed — Not Receiving any Study Medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants including one participant who was assigned to the UFH/Warfarin group and withdrew from the study prior to receiving any study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (13.40) | 66.1 (17.72) | 65.2 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 22 | 17 | 39
Primary Diagnosis, Deep Venous Thrombosis (DVT)/Pulmonary Embolism (PE) [Number; unit: participants]
  DVT | 22 | 23 | 45
  PE | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Bleeding Events ［Per International Society on Thrombosis and Homeostasis (ISTH) Definition］ or Clinically Relevant Non-major (CRNM) Bleeding Events Adjudicated by Clinical Event Committee During the Treatment Period
Description: Major bleeding event was defined as an acute clinically overt bleeding accompanied by a decrease in hemoglobin of 2 g/dL or more, a transfusion of 4 or more units of packed red blood cells (a unit of packed red blood cells equal to about 200 cc), or bleeding that occurred in critical sites (e.g. intracranial). Fatal bleeding was also defined as a major bleeding event. CRNM bleeding event was defined as an acute clinically overt bleeding that did not satisfy the definition of major bleeding and that led to either hospitalization, physician guided medical or surgical treatment for bleeding, or a change in antithrombotic therapy.
Time Frame: Baseline to Week 24
Population: The safety analysis set (SAS) consisted of all treated participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 40 | 39
participants | 3 | 11

2. Secondary Outcome: Number of Participants With Adjudicated Recurrent Symptomatic Venous Thromboembolism (VTE) ［Nonfatal Deep Venous Thrombosis (DVT) or Nonfatal Pulmonary Embolism (PE)］ or VTE-Related Death During the Intended Treatment Period
Description: VTE-related death was defined as a death caused by documented PE which was diagnosed with objective testing or autopsy, or an unexplained death for which DVT/PE could not be ruled out as the cause. "Intended Treatment Period" was the period starting on the day of randomization and ending at either 2 days after the last dose of the study drug or Day 168/Week 24, whichever came late.
Time Frame: Baseline to Week 24
Population: Full analysis set (FAS) was defined as all randomized participants. Participants with missing endpoint information were excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 38 | 40
participants | 0 | 1

3. Secondary Outcome: Number of Participants With Adjudicated Thrombotic Burden Worsened in Acute Symptomatic Proximal Deep Venous Thrombosis (DVT)
Description: Computed tomography venography (CTV) and compression ultrasound (CUS) were used to assess thrombotic burden in the participants with DVT and the results were classified as improved, no change, or worsened. The timings of CTV and CUS examinations were at Week 12 and Weeks 2, 12 and 24.
Time Frame: Baseline to Week 24
Population: A subset of full analysis set (FAS) that consisted of participants with DVT. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 22 | 23
participants
  CUS - Week 2 (n=22, n=22) | 1 | 2
  CTV - Week 12 (n=20, n=21) | 0 | 0
  CUS - Week 12 (n=21, n=22) | 0 | 0
  CUS - Week 24 (n=20, n=22) | 0 | 1

4. Secondary Outcome: Number of Participants With Adjudicated Thrombotic Burden Worsened in Acute Symptomatic Pulmonary Embolism (PE)
Description: Computed tomography pulmonary angiography (CTPA) was used to assess thrombotic burden in the participants with PE and the results were classified as improved, no change, or worsened. The timings of CTPA examinations were Weeks 2, 12 and 24.
Time Frame: Baseline to Week 24
Population: A subset of full analysis set (FAS) that consisted of participants with PE. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 18 | 17
participants
  CTPA - Week 2 (n=18, n=17) | 0 | 0
  CTPA - Week 12 (n=18, n=16) | 0 | 0
  CTPA - Week 24 (n=16, n=15) | 0 | 1

5. Secondary Outcome: Number of Participants With Adjudicated Major Bleeding Events ［Per International Society on Thrombosis and Homeostasis (ISTH) Definition］During the Treatment Period
Description: Major bleeding event was defined as an acute clinically overt bleeding accompanied by a decrease in hemoglobin of 2 g/dL or more, a transfusion of 4 or more units of packed red blood cells (a unit of packed red blood cells equal to about 200 cc), or bleeding that occurred in critical sites (e.g. intracranial). Fatal bleeding was also defined as a major bleeding event.
Time Frame: Baseline to Week 24
Population: The safety analysis set (SAS) consisted of all treated participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 40 | 39
participants | 0 | 2

6. Secondary Outcome: Number of Participants With Adjudicated All Bleeding Events During the Treatment Periods
Description: All bleeding events consisted of major bleeding (per Interactional Society on Thrombosis and Homeostasis ［ISTH］ Definition), clinically relevant non-major (CRNM) and minor bleeding. All acute clinically overt bleeding events not meeting the criteria for either major bleeding or CRMN bleeding were classified as minor bleeding.
Time Frame: Baseline to Week 24
Population: The safety analysis set (SAS) consisted of all treated participants.
Measure: Number; unit: participants
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Number analyzed (Participants) | 40 | 39
participants | 7 | 17

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what are presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Apixaban | Unfractionated Heparin (UFH)/Warfarin
Serious Adverse Events (participants affected / at risk) | 3/40 | 7/39
Other Adverse Events (participants affected / at risk) | 29/40 | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Apixaban (N=40) | Unfractionated Heparin (UFH)/Warfarin (N=39)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0/4 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=40) | Unfractionated Heparin (UFH)/Warfarin (N=39)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 4 | 5
Bronchopneumonia (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 4 | 4
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood triglycerides increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 5
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.